CLINICAL TRIAL: NCT02379208
Title: Evaluation of Rate of Progression With Perimetry in Newly Diagnosed Open Angle Glaucoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: T58/2012
Record Dates: First submitted 2015-02-03; First posted 2015-03-04 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-02

CONDITIONS: Glaucoma, Open-Angle; Ocular Hypertension
Keywords: Visual Field Tests; Ocular Hypertension; Glaucoma, Open-Angle; Quality of Life; Glaucoma progression; Early glaucoma; Frequency Doubling Technology (FDT); RareBit; Octopus 900 perimetry
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Glaucoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to evaluate rate of progression in newly diagnosed open angle glaucoma with different types of perimetry. Would it be possible to find the rapidly progressing individuals sooner by doing perimetry more often? Is there a difference between different types of perimetry in early glaucoma? What would be the optimal timing of perimetry in newly diagnosed glaucoma? In addition the quality of life in glaucoma patients will be evaluated with two types of questionnaires in three different time points. The enrolled patients will receive appropriate treatment according to glaucoma management guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed open angle glaucoma

Exclusion Criteria:

* Significant visual impairment due to another disease (e.g. diabetic retinopathy or maculopathy, cataract, visual field defect after stroke)
* Inability to perform perimetry reliably

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients referred to Turku University Central Hospital for suspected or newly diagnosed open angle glaucoma
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2015-04; Primary Completion 2019-12 (Estimated); Study Completion 2020-05 (Estimated)

PRIMARY OUTCOMES:
Change in mean defect in Octopus perimetry | Baseline, 2, 4, 8, 12, 16, 20, 22, 24 months

SECONDARY OUTCOMES:
Change in VF-7- instrument score | 2, 12, 24 months
  Change in quality of life
Change in 15D-instrument score | 2, 12, 24 months
  Change in quality of life
Differences in visual field defects between Octopus, frequency doubling technology, RareBit-perimeters | 2, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Eija Vesti, Professor, Study Director — University of Turku
Locations (1):
- Turku University Central Hospital, Turku, Finland